CLINICAL TRIAL: NCT00460161
Title: Acupuncture for Phantom Limb Pain: A Randomized, Double-Blind, Placebo/Sham - Controlled Study
Brief Title: Acupuncture for Phantom Limb Pain
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Noah Samuels, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACP.PLP.10.06
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2008-08

CONDITIONS: Phantom Limb Pain
Keywords: acupuncture; amputation; phantom limb pain
MeSH Terms: conditions — Phantom Limb | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): true acupuncture
  Interventions: Procedure: acupuncture
- 2 (Placebo Comparator): placebo/sham acupuncture
  Interventions: Other: placebo/sham acupuncture

INTERVENTIONS:
Procedure: acupuncture — 2 treatments/week for 4 weeks
  Arms: 1
Other: placebo/sham acupuncture — 2 treatments/week for 4 weeks
  Arms: 2

SUMMARY:
Phantom pain is a common complication following limb amputation, and is thought to result from a system of pathophysiological mechanisms - peripheral, spinal, central and psychological. Treatment is primarily medical, using antidepressant and anticonvulsant medications. At present, there is no evidence-based approach for the management of phantom limb pain (PLP). Acupuncture is an ancient Chinese treatment during which thin needles (diameter 0.20-0.30mm) are inserted into various points on the skin. Studies of this treatment have found significant benefit in a number of conditions with chronic pain.

We propose a randomized, double-blind, placebo/sham -controlled study to evaluate whether acupuncture is an effective and safe modality for preventing and reducing PLP in patients following lower limb amputation. Patients requiring lower limb amputation (above-ankle) will be randomized into two groups, for real or placebo/sham acupuncture treatment. Both groups will be treated twice-weekly with a standardized (as opposed to individualized) acupuncture treatment protocol, using either true or placebo needles at sham acupuncture points, for a period of four weeks (eight treatments).

The primary outcome to be evaluated will be PLP at 4 weeks, using a site-specific numerical rating pain scale (ss-NRS). Secondary outcome measures to be evaluated are: stump pain (ss-NRS); analgesic use (Tramadol, 100mg Tablet); and depressive symptoms, using the Beck Depression Score. Blinding of the participants will be evaluated using a Validation of Blinding Questionnaire at the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender
* Age 18 years and older
* Scheduled for lower single limb amputation (above or below knee)
* Ability to comply with study protocol

Exclusion Criteria:

* Patients requiring limb amputation due to trauma
* Patients displaying symptoms of overt Axis-1 psychopathology such as Schizophrenia or Substance Abuse
* Inability to comply with the study protocol
* Previous experience with acupuncture treatment; current use of complementary or alternative medical treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
To study the effect of acupuncture on phantom limb pain at 4 weeks post-amputation | 4 weeks

SECONDARY OUTCOMES:
To study the effect of acupuncture on phantom limb pain at 3 months post-amputation | 3 months
To study the effect of acupuncture on stump pain at 4 weeks post-amputation | 4 weeks
To study the effect of acupuncture on analgesic use (Tramadol 100mg) during the first 4 weeks post-amputation | 4 weeks
To study the effect of acupuncture on parameters of depression (using the Beck Depression Score) at 4 weeks and 3 months post-amputation | 4 weeks and 3 months
To study the safety of acupuncture treatment in patients following amputation with phantom limb pain | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Noah Samuels, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel